CLINICAL TRIAL: NCT00655837
Title: A Phase Ib Study of SGN-40 in Combination With Rituximab and Gemcitabine for the Treatment of Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Trial to Define the Safety and Tolerability of SGN-40, Rituximab, and Gemcitabine in Patients With DLBCL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG040-0008
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin
Keywords: Antigens, CD40; Antibodies, Monoclonal; Combined Modality Therapy; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hematologic Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hematologic Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Lymphoma | interventions — dacetuzumab; Rituximab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SGN-40; Drug: rituximab; Drug: gemcitabine

INTERVENTIONS:
Drug: SGN-40 — 4-12mg/kg IV; Days 1, 4, 8, 15 and 22 of Cycle 1 and Days 1, 8 and 15 of Cycles 2-8.
  Other Names: dacetuzumab
Drug: rituximab — 375 mg/m2 IV injection; Days -2, 8, 15 and 22 of Cycle 1 and Day 1 of Cycles 2-8.
  Other Names: Rituxan
Drug: gemcitabine — 1000 mg/m2 IV Injection; Days 1 and 15 of all Cycles.
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to determine safety and tolerability of combination therapy of SGN-40 with gemcitabine and rituximab for the treatment of lymphoma. This study is also intended to estimate how well your disease responds to this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologic diagnosis of DLBCL, including transformed histology and follicular grade 3 disease.
* Must have at least one site of biopsy-proven disease demonstrating both of the following: bidimensional measurable disease with the longest axis >= 1.5cm by radiographic imaging or positive FDG-PET scan at baseline.
* Patients with DLBCL and who have either relapsed, refractory, or progressive disease following salvage therapy, OR relapsed, refractory, or progressive disease following initial therapy and be medically unfit to receive aggressive therapy.
* Either fresh or archived tumor specimen must be available.

Exclusion Criteria:

* Documented history within 6 months of registration of a cerebral vascular event, unstable angina, myocardial infarction, or cardiac symptoms.
* Patients who have received allogeneic stem cell transplant.
* Patients with evidence of another invasive primary malignancy within the past three years other than non-melanoma skin cancer, cervical carcinoma in situ, in situ carcinoma of the breast, or fully resected prostate cancer with normal PSA within 8 weeks of registration.
* Patients with any active systemic viral, bacterial, or fungal infection requiring intravenous anti-infectives within 4 weeks prior to first dose of study drug.
* Patients with a history or clinical evidence of leptomeningeal or central nervous system (CNS) lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Determine the safety and adverse-event profile for combination therapy of SGN-40 with gemcitabine and rituximab. | 10 months from registration of last patient

SECONDARY OUTCOMES:
Estimate progression free survival, clinical response rates to treatment, and overall survival to determine efficacy. | Follow-up every 6 weeks after end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Whiting, PharmD, Study Director — Seagen Inc.
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of Colorado, Aurora, Colorado
  - Oncology Specialists, Park Ridge, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Forero-Torres A, Bartlett N, Beaven A, Myint H, Nasta S, Northfelt DW, Whiting NC, Drachman JG, Lobuglio AF, Moskowitz CH. Pilot study of dacetuzumab in combination with rituximab and gemcitabine for relapsed or refractory diffuse large B-cell lymphoma. Leuk Lymphoma. 2013 Feb;54(2):277-83. doi: 10.3109/10428194.2012.710328. Epub 2012 Sep 8. PMID 22775314